CLINICAL TRIAL: NCT05373732
Title: Stress Reduction in the Prevention of Left Ventricular Hypertrophy: A Randomized Controlled Trial of Transcendental Meditation and Health Education in Hypertensive African Americans
Brief Title: Stress Reduction in the Prevention of Left Ventricular Hypertrophy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maharishi International University (Other)
Collaborators: Charles Drew University of Medicine and Science (Other)
Responsible Party: Principal Investigator, Robert Schneider, MD, Director and Dean, Maharishi International University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2100mdmvc
Record Dates: First submitted 2022-04-06; First posted 2022-05-13 (Actual); Last update posted 2022-05-13 (Actual); Status verified 2022-05

CONDITIONS: Left Ventricular Hypertrophy; High Blood Pressure
Keywords: left ventricular mass; meditation; stress reduction
MeSH Terms: conditions — Hypertrophy, Left Ventricular; Hypertension | interventions — Meditation; Mindfulness-Based Stress Reduction

STUDY DESIGN:
Intervention Model Description: A randomized, controlled, single-blinded, clinical trial was conducted to compare the effect of Transcendental Meditation (TM) and health education (HE) on left ventricular mass in adult hypertensive African-Americans
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomization was stratified by age, gender, mean arterial pressure, left ventricular mass index (LVMI), and antihypertensive medication. Investigators, data collectors and data management staff were blinded to group assignment. The biostatistician concealed the allocation by conveying the group assignment to the project manager who then informed each participant and instructed them not to reveal it to the research and data collection staff during the course of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transcendental Meditation (Experimental): The Transcendental Meditation (TM) technique is described as a simple, natural technique that is practiced twice a day for 20 minutes while sitting comfortably with eyes closed. There are no required changes in lifestyle, beliefs or philosophy. Instruction in the TM technique involves a seven-step course over five sessions (90-minute meetings).
  Interventions: Behavioral: meditation
- Health Education (Active Comparator): The health education (HE) intervention provided behavioral instructions for CVD risk factor prevention . This group received written materials, structured presentations, didactic instructions and group support for modifying the major cardiovascular risk factors including salt restriction, weight reduction, aerobic exercise, alcohol and smoking cessation.
  Interventions: Behavioral: Health education control

INTERVENTIONS:
Behavioral: meditation — meditation practice 20 minutes twice a day at home and attending classes at the clinic.
  Other Names: stress reduction
  Arms: Transcendental Meditation
Behavioral: Health education control — didactic based classes in CVD risk factor reduction and prevention
  Arms: Health Education

SUMMARY:
This study evaluated the effect of stress reduction by Transcendental Meditation (TM) on left ventricular mass compared to a health education control group in pre-hypertensive or hypertensive African-American adults over a six-month intervention period.

DETAILED DESCRIPTION:
Left ventricular hypertrophy (LVH) is an independent risk factor for cardiovascular disease (CVD). African Americans have higher rates of LVH and CVD than whites. Substantial evidence indicates that psychological stress contributes to LVH. This randomized controlled trial evaluated the effect of stress reduction with the Transcendental Meditation (TM) technique on left ventricular mass (LVM) in hypertensive African-Americans.

Hypertensive African American men and women were tested at baseline for left ventricular mass index (LVMI) by M-mode echocardiography, blood pressure, lifestyle and behavioral factors. Subjects were randomly assigned to either TM or health education (HE) control. After six months intervention, 86 subjects were posttested on all outcomes. Data were analyzed for between-group and within-group differences.

ELIGIBILITY:
Inclusion Criteria: self-identified African-American men and women ages, 20-75 years old, with either prehypertension (systolic blood pressure (SBP) of 120-139 mm Hg and/or diastolic blood pressure (DBP) of 80-89 mm Hg), Stage-1 hypertension (SBP of 140-159 mm Hg and/or DBP of 90-99 mm Hg) or Stage-2 hypertension (SBP of 160-179 and/or DBP of 100-109 mm of Hg), with or without antihypertensive medications -

Exclusion Criteria: Patients with a history of stroke, transient cerebral ischemic attack, congestive heart failure, myocardial infarction, angina pectoris or with significant ECG abnormalities, major psychiatric or behavioral disorder such as alcoholism (> 28 drinks per week)

-

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 1996-04 (Actual); Primary Completion 1998-10 (Actual); Study Completion 1998-12 (Actual)

PRIMARY OUTCOMES:
left ventricular mass (LVM) | 6 months pre to post
  The primary outcome was change in LVMI. LVM was measured by M-mode echocardiography and indexed by body surface area to generate LVMI. [18] Measurements were obtained at the end-diastole. Interventricular septal thickness, posterior wall thickness, and left ventricle internal dimension were measured.

SECONDARY OUTCOMES:
blood pressure | 0 and 6 months
  systolic and diastolic blood pressure
anger expression | 0 and 6 months
  Speilberger Anger expression scale
perceived stress | 0 and 6 months
  Perceived Stress Scale, a 5-item subset of the California Self-Evaluation Scale to measure self-esteem, and a personal efficacy scale

CONTACTS AND LOCATIONS:
Overall Officials: Robert H Schneider, M.D., Principal Investigator — Maharishi International University

IPD SHARING:
Plan to Share IPD: Yes
IPD is available on request to authors from other study investigators. Database on Excel is available to be emailed to inquiring investigators
Supporting Information: Study Protocol, SAP, ICF
Time Frame: currently available
Access Criteria: contact investigators and request access to database and submit short study proposal

REFERENCES:
- [Result] Schneider RH, Myers HF, Marwaha K, Rainforth MA, Salerno JW, Nidich SI, Gaylord-King C, Alexander CN, Norris KC. Stress Reduction in the Prevention of Left Ventricular Hypertrophy: A Randomized Controlled Trial of Transcendental Meditation and Health Education in Hypertensive African Americans. Ethn Dis. 2019 Oct 17;29(4):577-586. doi: 10.18865/ed.29.4.577. eCollection 2019 Fall. PMID 31641325